CLINICAL TRIAL: NCT03848871
Title: The Effect of Enstilar Versus Vehicle on Target Lesions in Moderate Plaque Type Psoriasis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research, PLLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENS-1702
Record Dates: First submitted 2019-02-06; First posted 2019-02-21 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enstilar foam (Experimental): Subjects will receive calcipotriene hydrate/betamethasone dipropionate (Enstilar) foam and apply to affected areas once daily. A target lesion located on elbow or knee will be identified by the Investigator for daily treatment with the medicated foam from Baseline through week 4.
  Interventions: Drug: Enstilar

INTERVENTIONS:
Drug: Enstilar — Enstilar foam applied to affected area once daily
  Other Names: calcipotriene and betamethasone dipropionate

SUMMARY:
This study seeks to show whether there is a benefit of prescribing Enstilar in the treatment of patients with moderate plaque type psoriasis. Subjects will receive study treatment of Enstilar foam.

DETAILED DESCRIPTION:
Approximately 20 subjects from 3 sites will be enrolled in this open-label study. Subjects will receive Enstilar foam and all adverse events and concomitant medications will be recorded.

Subjects will attend a screening visit/baseline visit and those with plaque-type psoriasis and bilateral symmetric psoriatic plaques will have a target lesion identified on knees or elbows and subjects will receive study treatment as outlined above.

Enstilar will be initiated daily for the entire study period of four weeks. Study visits will occur as follows: screening/baseline, week 2, week 4. Study assessments at each visit will be Body Surface Area (BSA,) Physicians Global Assessment (PGA,) Target lesion size, Total Lesion Severity Score (TLSS) and standard medical assessments. There will be standard medication/treatment and washout periods.

NOTE: The original study protocol dated december 20, 2017, was designed to compare the effect of Enstilar versus vehicle for the treatment of plaque psoriasis at a 1:1 ratio. A protocol amendment on March 20, 2018 eliminated the chance of placebo and made this an open-label study of the effects of Enstilar for the treatment of plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female subjects of any race, 18 years of age or higher. Female subjects of childbearing potential must have a (-) urine pregnancy test (UPT) result within 7 days of the first dose of study drug and practice a reliable method of contraception throughout the study.

   A female is considered of childbearing potential unless she is:

   - postmenopausal >5 years, without a uterus and/or both ovaries, or has been surgically sterile for >6 months

   Reliable methods of contraception are:

   - hormonal methods or intrauterine device (IUD) in use > 90 days prior to study drug administration, barrier methods plus spermicide in use > 14 days prior, or vasectomized partner.

   [Exception: Female subjects of child bearing potential (CBP) who are not sexually active are not required to practice a reliable method of contraception and may be enrolled at the Investigator's discretion provided they are counselled to remain sexually inactive for the duration of the study and understand the risks involved in getting pregnant during the study.]
2. Moderate plaque type psoriasis eligible for topical therapies.
3. Patients with a minimum of 3% BSA to a maximum of 20% BSA & bilateral symmetric psoriatic plaques of 2 to 4 cm in diameter.
4. Physician Global Assessment (PGA) score of 3.
5. Able to understand study requirements and sign Informed Consent/HIPAA forms.

   -

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control, or male subjects planning a pregnancy with their spouse or partner while in the study.
2. History of hypercalcaemia or vitamin D toxicity.
3. Patients with guttate, erythrodermic, or pustular psoriasis
4. Serious skin condition (other than psoriasis) or uncontrolled medical condition (in the opinion of the investigator.)
5. Topical steroids, topical immunomodulators, topical vitamin D derivatives, tar, salicylic acid, anthralin or any other topical treatment for psoriasis within 2 weeks of baseline.
6. Use of any biologics within 3 months of baseline.
7. Use of other systemic psoriasis treatments (ie, oral retinoids, methotrexate, cyclosporine, or other immunomodulators) within 4 weeks of baseline.
8. Use of ultraviolet B rays (UVB) or psoralen+ultraviolet a rays (PUVA) within 2 weeks of baseline.
9. Skin conditions (e.g. eczema) other than psoriasis that may interfere with evaluations of psoriasis.
10. Known hypersensitivity to Enstilar or any of its components.
11. Contraindications according to Enstilar.
12. Current drug or alcohol abuse (Investigator opinion.)
13. Subject unable to commit to all the assessments required by protocol. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DermResearch, PLLC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enstilar Foam
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Physicians Global Assessment (PGA) From Baseline to Week 2 and Week 4
Description: Physician assessment of disease severity. 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate
Time Frame: screening/baseline, week 2, week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 20
Participants
  Baseline: Moderate | 20
  Baseline: Mild | 0
  Baseline: Almost Clear | 0
  Baseline: Clear | 0
  Week 2: Moderate | 1
  Week 2: Mild | 13
  Week 2: Almost Clear | 6
  Week 2: Clear | 0
  Week 4: Moderate | 1
  Week 4: Mild | 4
  Week 4: Almost Clear | 9
  Week 4: Clear | 6

2. Secondary Outcome: Change in Lesion Size From Baseline to Week 2 and Week 4
Description: Size of target lesion recorded as height in cm x length in cm
Time Frame: screening/baseline, week 2, week 4
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 20
cm^2
  Baseline | 19 (14)
  Week 2 | 16 (13)
  Week 4 | 10 (8)

3. Secondary Outcome: Change in Body Surface Area (BSA) From Baseline to Week 2 and Week 4
Description: Percent of total body surface affected by psoriasis, calculated by multiplying the percent of a specified body area affected by psoriasis x the percent of total body surface area represented by the specified area (where head = 10% of total body surface, trunk = 30%, upper limbs = 20%, lower limbs = 40%)
Time Frame: screening/baseline, week 2, week 4
Measure: Mean (Standard Deviation); unit: percentage of body covered by psoriasis
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 20
percentage of body covered by psoriasis
  Baseline | 9.8 (6.8)
  Week 2 | 9.2 (6.9)
  Week 4 | 6.9 (7.5)

4. Secondary Outcome: Change in TLSS (Total Lesion Severity Score) From Baseline to Week 2 and Week 4 - Assessment of Erythema
Description: A combined score of disease severity of target lesion which includes assessment of erythema (0=none, 1= slightly pink, 2=pink, 4=red, 6=very red, 8=extremely red), induration (0=no evidence of plaque above normal skin level, 2=slight definite elevation above normal skin level, 4=moderate elevation with rounded or sloped edges to plaque, 6=marked elevation with hard sharp edges to plaque), and scaling (0=no evidence of scaling on lesion, 2= mild mainly fine scales with some of lesion at least partially covered, 4=moderate somewhat coarser scale and most of lesion at least partially covered, 6= severe coarse thick scales and rough surface covering virtually all of lesion, 8=very severe coarse very thick scales and rough surface covering entire lesion
Time Frame: screening/baseline, week 2, week 4
Population: Erythema assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 20
Participants
  Baseline: 8 Extremely Red | 0
  Baseline: 6 Very Red | 5
  Baseline: 4 Red | 13
  Baseline: 2 Pink | 2
  Baseline: 1 Slightly Pink | 0
  Baseline: 0 None | 0
  Week 2: 8 Extremely Red | 0
  Week 2: 6 Very Red | 0
  Week 2: 4 Red | 4
  Week 2: 2 Pink | 14
  Week 2: 1 Slightly Pink | 1
  Week 2: 0 None | 1
  Week 4: 8 Extremely Red | 0
  Week 4: 6 Very Red | 0
  Week 4: 4 Red | 4
  Week 4: 2 Pink | 7
  Week 4: 1 Slightly Pink | 1
  Week 4: 0 None | 8

5. Secondary Outcome: Change in TLSS (Total Lesion Severity Score) From Baseline to Week 2 and Week 4 - Assessment of Induration
Description: A combined score of disease severity of target lesion which includes assessment of erythema (0=none, 2=pink, 4=red, 6=very red, 8=extremely red), induration (0=no evidence of plaque above normal skin level, 1=very slight, 2=slight definite elevation above normal skin level, 3=mild, 4=moderate elevation with rounded or sloped edges to plaque, 6=marked elevation with hard sharp edges to plaque), and scaling (0=no evidence of scaling on lesion, 2= mild mainly fine scales with some of lesion at least partially covered, 4=moderate somewhat coarser scale and most of lesion at least partially covered, 6= severe coarse thick scales and rough surface covering virtually all of lesion, 8=very severe coarse very thick scales and rough surface covering entire lesion
Time Frame: screening/baseline, week 2, week 4
Population: Induration assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 20
Participants
  Baseline: 6 Marked | 5
  Baseline: 4 Moderate | 13
  Baseline: 3 Mild | 0
  Baseline: 2 Slight | 2
  Baseline: 1 Very Slight | 0
  Baseline: 0 None | 0
  Week 2: 6 Marked | 0
  Week 2: 4 Moderate | 3
  Week 2: 3 Mild | 1
  Week 2: 2 Slight | 9
  Week 2: 1 Very Slight | 1
  Week 2: 0 None | 6
  Week 4: 6 Marked | 0
  Week 4: 4 Moderate | 0
  Week 4: 3 Mild | 0
  Week 4: 2 Slight | 8
  Week 4: 1 Very Slight | 1
  Week 4: 0 None | 11

6. Secondary Outcome: Change in TLSS (Total Lesion Severity Score) From Baseline to Week 2 and Week 4 - Assessment of Scaling
Description: A combined score of disease severity of target lesion which includes assessment of erythema (0=none, 2=pink, 4=red, 6=very red, 8=extremely red), induration (0=no evidence of plaque above normal skin level, 2=slight definite elevation above normal skin level, 4=moderate elevation with rounded or sloped edges to plaque, 6=marked elevation with hard sharp edges to plaque, 8=very marked elevation with very hard sharp edges to plaque), and scaling (0=no evidence of scaling on lesion, 2= mild mainly fine scales with some of lesion at least partially covered, 4=moderate somewhat coarser scale and most of lesion at least partially covered, 6= severe coarse thick scales and rough surface covering virtually all of lesion, 8=very severe coarse very thick scales and rough surface covering entire lesion)
Time Frame: screening/baseline, week 2, week 4
Population: Scaling assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Enstilar Foam
Number analyzed (Participants) | 20
Participants
  Baseline: 8 Very Severe | 0
  Baseline: 6 Severe | 7
  Baseline: 4 Moderate | 12
  Baseline: 2 Mild | 1
  Baseline: 0 None | 0
  Week 2: 8 Very Severe | 0
  Week 2: 6 Severe | 0
  Week 2: 4 Moderate | 1
  Week 2: 2 Mild | 10
  Week 2: 0 None | 9
  Week 4: 8 Very Severe | 0
  Week 4: 6 Severe | 0
  Week 4: 4 Moderate | 1
  Week 4: 2 Mild | 4
  Week 4: 0 None | 15

ADVERSE EVENTS:
Time Frame: 4 weeks average, from signing of Informed consent until end of study participation
Arm/Group | Enstilar Foam
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enstilar Foam (N=20)
GERD exacerbation (Gastrointestinal disorders) | 1 (1)
dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT03848871/Prot_SAP_000.pdf